CLINICAL TRIAL: NCT04854174
Title: An Open-Label Food Effect Study of ZN-d5 in Healthy Female Volunteers
Brief Title: A Food Effect Study of ZN-d5 in Healthy Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: K-Group Alpha, Inc., a wholly owned subsidiary of Zentalis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZN-d5-002
Record Dates: First submitted 2021-03-17; First posted 2021-04-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteer (Experimental): Healthy Volunteer
  Interventions: Drug: ZN-d5

INTERVENTIONS:
Drug: ZN-d5 — Oral agent; 25 mg formulation
  Other Names: Study Drug

SUMMARY:
This is a single-center, sequential, open-label, food effect study to determine the comparative bioavailability of ZN-d5 under fasting and fed conditions, following single-dose oral administration of ZN-d5. The study will be comprised of a pre-study screening, followed by administration of a single dose of ZN-d5 under fasted conditions, a washout period, administration of a single dose of ZN-d5 under fed conditions, and a follow-up period.

DETAILED DESCRIPTION:
This is a single-center, sequential, open-label, food effect study to determine the comparative bioavailability of ZN-d5 under fasting and fed conditions, following single-dose oral administration of ZN-d5. The study will be comprised of a pre-study screening, followed by administration of a single dose of ZN-d5 under fasted conditions, a washout period, administration of a single dose of ZN-d5 under fed conditions, and a follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy females, age 18-65 years;
2. Body mass index (BMI) ≥ 18.0 and ≤ 29.9 kg/m2 and weight ≥ 50 kg and ≤ 100 kg at Screening;
3. Non-smoker and must not have used any tobacco products within two months prior to Screening, or if a smoker, must be currently (and for the last two months prior to screening) smoking ≤ 2 cigarettes or equivalent per week. Participants must be willing to abstain from the use of tobacco and products containing nicotine from 14 days prior to administration of study drug for the duration of the study;
4. No relevant dietary restrictions; willing to consume a high calorie, high fat breakfast and other standard meals provided during the domiciled periods of the study, to comply with the fasting conditions required by the study design, and to avoid consumption of grapefruit, carambola (star fruit), pomelo or Seville oranges or their juices or extracts from 7 days prior to the administration of study drug and for the duration of the study;
5. Willing to abstain from alcohol beginning 48 hours prior to each admission until discharge from the study center at the end of each domiciled period;
6. Able to take and retain oral medications;
7. If sexually active and of childbearing potential, must agree to use two effective methods of contraception beginning at the Screening Visit until 60 days following the last dose of study drug; egg donation is also prohibited during this period (see Appendix 14.1). Post-menopausal status to be confirmed with serum follicle-stimulating hormone (FSH) levels;
8. Negative serum pregnancy test; i.e., beta-human chorionic gonadotropin (β-hCG) test at Screening and negative urine pregnancy test prior to administration of study drug (unless post-menopausal status is FSH-confirmed);
9. Must have the ability and willingness to attend the necessary visits to the study center and to be domiciled overnight where required;
10. Provides written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures;
11. Baseline B lymphocyte count >150 cells/µL (0.15 x109 cells/L).

Exclusion Criteria:

1. Any condition possibly affecting drug absorption (e.g., gastrectomy, gastric banding, or gastric bypass);
2. Prior or ongoing medical conditions, medical history, physical findings, or laboratory abnormality that, in the Investigator's opinion, could adversely affect the safety of the participant or make it unlikely that the participant will comply with the protocol or complete the study per protocol;
3. Blood donation or significant blood loss within 60 days prior to the first study drug administration or plasma donation within 7 days of the administration of study drug;
4. Routine consumption of xanthine-containing products or foods exceeds 800 mg daily intake of xanthines, continuing to within 7 days of the administration of study drug;
5. Fever (body temperature ≥38°C) or symptomatic viral or bacterial infection or febrile illness within 2 weeks prior to Screening;
6. History of recurrent (more than three episodes in 12 months) or chronic infections of any type, such as tuberculosis, sinusitis, or urinary tract infection, that in the opinion of the Investigator poses a risk to participate in the study, or any infection requiring parenteral antibiotics within the six months prior to Screening;
7. 12-lead ECG demonstrating QT interval corrected for heart rate using Fridericia's formula (QTcF) > 480 msec at the Screening Visit or history/evidence of long QT syndrome;
8. Other abnormal ECG findings at Screening that are considered by the investigator to be clinically significant;
9. Alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), and/or total bilirubin > 1.5 × upper limit of normal at screening (elevated bilirubin acceptable if participant was known to have Gilbert's syndrome). Repeat testing at Screening is acceptable for out-of-range values following approval by the Investigator or delegate;
10. Estimated glomerular filtration rate by CKD-EPI <60 mL/min/1.73 m2
11. Pregnant or breast-feeding, or intending to become pregnant, initiate breast-feeding or donate eggs from Screening until 60 days after the last dose of study drug;
12. Positive serology test for hepatitis C antibody (HCV), hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) antibody at Screening;
13. Positive urine toxicology screening panel or alcohol breath test;
14. History of substance abuse or dependency or history of recreational intravenous drug use over the last 5 years (by self-declaration);
15. Regular alcohol consumption within the 6 months prior to study drug administration, defined as >14 alcohol units per week (where 1 unit = 284 mL of beer, 25 mL of 40% spirit or a 125 mL glass of wine);
16. Use of any investigational product within the longer of 28 days or 5 half-lives prior to administration of study drug or participation in more than four investigational drug studies within 1 year prior to Screening;
17. Use of any prescription drugs, over-the-counter (OTC) (non-prescription) medication, herbal remedies (including St John's Wort), supplements or vitamins 14 days prior to dosing and during the course of study without prior approval of the Investigator and Sponsor.

    Simple analgesia (e.g., paracetamol or OTC nonsteroidal anti-inflammatory drugs) are permitted in limited doses;
18. Use of strong or moderate inhibitors or inducers of Cytochrome P450 (CYP) 3A, inhibitors or inducers of P-glycoprotein (P-gp), or drugs known to prolong the QT interval during the longer of 14 days or five half-lives prior to enrollment and during the course of the study;
19. Unwilling or unable to comply with the lifestyle guidelines outlined in the protocol.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2021-06-13 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
ZN-d5 Bioavailability | 2 months
  Maximum concentration (Cmax)
ZN-d5 Bioavailability | 2 months
  Area under the plasma concentration-time curve (AUC)

SECONDARY OUTCOMES:
Safety and Tolerability of ZN-d5 | 2 Months
  The incidence, frequency and severity of treatment-emergent adverse events (TEAEs)
Safety and Tolerability of ZN-d5 | 2 months
  time to maximum concentration
Safety and Tolerability of ZN-d5 | 2 Months
  delay in achieving Tmax (tlag)
Safety and Tolerability of ZN-d5 | 2 Months
  Half-life (t1/2)
Safety and Tolerability of ZN-d5 | 2 months
  Volume of distribution (Vs/F)
Safety and Tolerability of ZN-d5 | 2 months
  Clearance (CL/F)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Fiorino, MD, PhD, Study Director — K-Group Alpha, Inc., a wholly owned subsidiary of Zentalis Pharmaceuticals, Inc.
Locations (1):
- Site # 2801, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No